CLINICAL TRIAL: NCT05688137
Title: Abdominal Drainage in the Postoperative Period of Liver Transplantation (DRALIT): Multi-institutional Randomized Clinical Trial
Brief Title: Abdominal Drainage in the Postoperative Period of Liver Transplantation (DRALIT)
Acronym: DRALIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Alvaro Cerezuela Fernandez de Palencia, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-3-9-HCUVA
Record Dates: First submitted 2022-05-31; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Liver Transplant; Complications; Drainage

STUDY DESIGN:
Intervention Model Description: 2 groups of equal size, total n = 365 patients. Simple intraoperative randomization prior to closure of the abdominal wall after fulfilling all the inclusion criteria and none of the exclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRAINAGE GROUP (D) (Active Comparator): This patients will take the abdominal drainage.
  Interventions: Procedure: Abdominal drainage
- NON DRAINAGE GROUP (ND) (No Intervention): This patients will not take the abdominal drainage.

INTERVENTIONS:
Procedure: Abdominal drainage — The patients with intervention will take an abdominal drainage.
  Arms: DRAINAGE GROUP (D)

SUMMARY:
Classically, in the postoperative period of liver transplantation (LT), abdominal drainage has been used as a way to make the early diagnosis of hemorrhages, bile leaks and other postsurgical complications, as well as an evacuation route for ascites. The use of it routinely is currently under discussion due to the morbidities associated with its use.

DETAILED DESCRIPTION:
LT has become in recent years a procedure with an increasing number of indications and with a greater number of donations given the social knowledge of the donation process and donation in controlled asystole. The Spanish Registry of Liver Transplantation (RETH) shows a total of 28,609 TH in the period 1986-2019, which represents an average of 867 TH per year in Spain. These data place Spain among the first countries in terms of HT.

In LT, abdominal drainage has historically been used prophylactically as a way to identify early intra-abdominal postoperative complications such as hemorrhage, bile leakage, and others.

In transplant patients, the use of post-surgical abdominal drains on a routine basis has shown an increase in total protein losses in patients with refractory ascites, an increase in ascending infections secondary to drainage, infection and pain at the insertion point of the drain, as well as as, an increase in hospital stay. Nor can a higher rate of postsurgical bleeding and bile leakage be ruled out in patients with abdominal drainage.

Currently, in the few studies that there are in reference to the systematic use of abdominal drains in lTH, the need for them prophylactically is being discussed as an early diagnosis of postoperative intra-abdominal complications is not observed, but complications are seen to increase secondary to drainage. Therefore, the need to use it systematically in all patients is currently under discussion.

Currently, is facing an increase in ERASⓇ (Enhanced Recovery After Surgey) programs, which began in 2008 with colorectal surgery and are currently expanding to other surgical procedures. These programs advocate reducing the number of drains and even not using them in patients with a low risk of post-surgical complications.

In the current bibliography, the methodology of the studies is varied, with the majority being non-randomized retrospective studies, which is why it is a subject that requires studies with a better methodological design and a higher number of patients to obtain conclusions of clinical relevance. that can set the direction in this area that is in constant discussion.

Given the absence of any randomized non-inferiority clinical trial that studies the routine use of abdominal drainage in the postoperative period of liver transplantation, consider that it is necessary to carry it out to increase the evidence.

The number of HT performed in each center is limited and variable annually, which is why consider that the best design for this clinical trial is a European multicenter.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged between 18 and 75 years included in the waiting list for HT by the committee of the Virgen de la Arrixaca University Hospital.
* Sign Informed Consent.

Exclusion Criteria:

* Having been rejected for liver transplantation by said committee.
* Age less than 18 years or greater than 75.
* Any contraindication by the main surgeon that makes the placement of an intra-abdominal drain necessary.
* Not having signed the Informed Consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal drainage complications | 90 days
  To assess whether the prophylactic use of abdominal drains in the postoperative period of LT increases the number of abdominal complications in the 90 postoperative days (Clavien-Dindo)

SECONDARY OUTCOMES:
Assessment of quality of life (QoL) during the perioperative process using the SF-36 questionnaire. | 120 days
  Assessment of the quality of life (QoL) of transplant recipients, whether or not they are drainage recipients, during the perioperative process using the SF-36 questionnaire.
Evaluation of in-hospital stay after surgery. | 90 days
  Evaluate the postoperative stay in both groups from the hospital admission to discharge measured in days of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Cerezuela Fernández de Palencia, Principal Investigator — Hospital Universitario Virgen de la Arrixaca

REFERENCES:
- [Background] Hobeika C, Cauchy F, Weiss E, Chopinet S, Sepulveda A, Dondero F, Khoy-Ear L, Grigoresco B, Dokmak S, Durand F, Le Roy B, Paugam-Burtz C, Soubrane O. Practical model to identify liver transplant recipients at low risk of postoperative haemorrhage, bile leakage and ascites. BJS Open. 2021 Jan 8;5(1):zraa031. doi: 10.1093/bjsopen/zraa031. PMID 33609380
- [Background] Schwarz C, Soliman T, Gyori G, Silberhumer G, Schoppmann SF, Muhlbacher F, Berlakovich GA. Abdominal drainage after liver transplantation from deceased donors. Langenbecks Arch Surg. 2015 Oct;400(7):813-9. doi: 10.1007/s00423-015-1338-3. Epub 2015 Sep 4. PMID 26341224
- [Background] Rodriguez-Laiz GP, Melgar-Requena P, Alcazar-Lopez CF, Franco-Campello M, Villodre-Tudela C, Pascual-Bartolome S, Bellot-Garcia P, Rodriguez-Soler M, Miralles-Macia CF, Mas-Serrano P, Navarro-Martinez JA, Martinez-Adsuar FJ, Gomez-Salinas L, Jaime-Sanchez FA, Perdiguero-Gil M, Diaz-Cuevas M, Palazon-Azorin JM, Such-Ronda J, Lluis-Casajuana F, Ramia-Angel JM. Fast-Track Liver Transplantation: Six-year Prospective Cohort Study with an Enhanced Recovery After Surgery (ERAS) Protocol. World J Surg. 2021 May;45(5):1262-1271. doi: 10.1007/s00268-021-05963-2. Epub 2021 Feb 23. PMID 33620540
- [Background] Gurusamy KS, Naik P, Davidson BR. Routine drainage for orthotopic liver transplantation. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD008399. doi: 10.1002/14651858.CD008399.pub2. PMID 21678376
- [Background] Arita J, Sakamaki K, Saiura A, Konishi M, Sakamoto Y, Hashimoto M, Sano T, Uesaka K, Kokudo N, Yamanaka T, Shimada K. Drain Placement After Uncomplicated Hepatic Resection Increases Severe Postoperative Complication Rate: A Japanese Multi-institutional Randomized Controlled Trial (ND-trial). Ann Surg. 2021 Feb 1;273(2):224-231. doi: 10.1097/SLA.0000000000004051. PMID 33064385
- [Background] Weiss S, Messner F, Huth M, Weissenbacher A, Denecke C, Aigner F, Brandl A, Dziodzio T, Sucher R, Boesmueller C, Oellinger R, Schneeberger S, Oefner D, Pratschke J, Biebl M. Impact of abdominal drainage systems on postoperative complication rates following liver transplantation. Eur J Med Res. 2015 Aug 21;20(1):66. doi: 10.1186/s40001-015-0163-z. PMID 26293656
- [Background] Brustia R, Monsel A, Skurzak S, Schiffer E, Carrier FM, Patrono D, Kaba A, Detry O, Malbouisson L, Andraus W, Vandenbroucke-Menu F, Biancofiore G, Kaido T, Compagnon P, Uemoto S, Rodriguez Laiz G, De Boer M, Orloff S, Melgar P, Buis C, Zeillemaker-Hoekstra M, Usher H, Reyntjens K, Baird E, Demartines N, Wigmore S, Scatton O. Guidelines for Perioperative Care for Liver Transplantation: Enhanced Recovery After Surgery (ERAS) Recommendations. Transplantation. 2022 Mar 1;106(3):552-561. doi: 10.1097/TP.0000000000003808. PMID 33966024
- [Background] Tang R, Yu LH, Han JW, Lin JY, An JJ, Lu Q. Abdominal drainage systems in modified piggyback orthotopic liver transplantation. Hepatobiliary Pancreat Dis Int. 2021 Feb;20(1):99-102. doi: 10.1016/j.hbpd.2020.09.003. Epub 2020 Sep 13. No abstract available. PMID 32967814
- [Background] Fernandez-Aguilar JL, Suarez Munoz MA, Santoyo Santoyo J, Sanchez-Perez B, Perez-Daga JA, Aranda Narvaez JM, Ramirez Plaza C, Becerra Ortiz R, Titos Garcia A, Gonzalez Sanchez A, Montiel Casado C. Is liver transplantation without abdominal drainage safe? Transplant Proc. 2010 Mar;42(2):647-8. doi: 10.1016/j.transproceed.2010.02.007. PMID 20304214
- [Background] Fernandez-Aguilar JL, Suarez-Munoz MA, Sanchez-Perez B, Gamez Cordoba E, Pulido Roa Y, Aranda Narvaez J, Perez Daga A, Montiel Casado C, Gonzalez Sanchez A, Santoyo Santoyo J. Liver transplantation without abdominal drainage. Transplant Proc. 2012 Nov;44(9):2542-4. doi: 10.1016/j.transproceed.2012.09.039. PMID 23146448
- [Background] Liu CL, Fan ST, Lo CM, Wong Y, Ng IO, Lam CM, Poon RT, Wong J. Abdominal drainage after hepatic resection is contraindicated in patients with chronic liver diseases. Ann Surg. 2004 Feb;239(2):194-201. doi: 10.1097/01.sla.0000109153.71725.8c. PMID 14745327
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Petrowsky H, Demartines N, Rousson V, Clavien PA. Evidence-based value of prophylactic drainage in gastrointestinal surgery: a systematic review and meta-analyses. Ann Surg. 2004 Dec;240(6):1074-84; discussion 1084-5. doi: 10.1097/01.sla.0000146149.17411.c5. PMID 15570212
- [Background] de Rougemont O, Dutkowski P, Weber M, Clavien PA. Abdominal drains in liver transplantation: useful tool or useless dogma? A matched case-control study. Liver Transpl. 2009 Jan;15(1):96-101. doi: 10.1002/lt.21676. PMID 19109839
- [Background] Sanada Y, Mizuta K, Urahashi T, Umehara M, Wakiya T, Okada N, Hayashida M, Egami S, Hishikawa S, Kawano Y, Ushijima K, Otomo S, Sakamoto K, Fujiwara T, Sakuma Y, Hyodo M, Yasuda Y, Kawarasaki H. Management of intra-abdominal drain after living donor liver transplantation. Transplant Proc. 2010 Dec;42(10):4555-9. doi: 10.1016/j.transproceed.2010.09.159. PMID 21168736
- [Background] Baldini E, Gugenheim J, Ouzan D, Katkhouda N, Mouiel J. Orthotopic liver transplantation with and without peritoneal drainage: a comparative study. Transplant Proc. 1999 Feb-Mar;31(1-2):556-7. doi: 10.1016/s0041-1345(98)01553-x. No abstract available. PMID 10083235
- [Background] Hampe T, Dogan A, Encke J, Mehrabi A, Schemmer P, Schmidt J, Stiehl A, Sauer P. Biliary complications after liver transplantation. Clin Transplant. 2006;20 Suppl 17:93-6. doi: 10.1111/j.1399-0012.2006.00607.x. PMID 17100708
- [Background] Thethy S, Thomson BNj, Pleass H, Wigmore SJ, Madhavan K, Akyol M, Forsythe JL, James Garden O. Management of biliary tract complications after orthotopic liver transplantation. Clin Transplant. 2004 Dec;18(6):647-53. doi: 10.1111/j.1399-0012.2004.00254.x. PMID 15516238

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT05688137/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT05688137/ICF_001.pdf